CLINICAL TRIAL: NCT06380465
Title: The Effect of Anthocyanin Intake From Purple Sweet Potato on Vasomotor Reactivity of Intracranial Vessels in Cerebral Small Vessel Disease - a Study of Breath-Holding Index, Nitric Oxide, L-Arginine, Adiponectin, Cognitive and Gait
Brief Title: The Effect of Anthocyanin Intake From Purple Sweet Potato in Cerebral Small Vessel Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); Universitas Padjadjaran (Other); Institut Pertanian Bogor (Other); School of Science and technology, Kwansei Gakuin University (Unknown)
Responsible Party: Principal Investigator, dr.Taufik Mesiano,Sp.S (K), Doctoral Program, Medical Staff & Lecturer, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-11-1838
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: anthocyanin; purple sweet potato; vasomotor reactivity; cerebral small vessel disease; BHI; nitric oxide; l-arginine; adiponectin; cognitive; gait
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Intervention Model Description: The participant who meet the inclusion criteria and have signed the consent will be subjected to a baseline assessment followed by randomization into 2 groups/arms consisting of 2 treatments (1 group getting the water extract pf purple sweet potato) and 1 control group that got placebo.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research was conducted using a single-blind approach, where the participants were unaware of the intervention being implemented
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1:1 water extract of purple sweet potato (Experimental): subjects were blindly and randomly assigned the pure water extract of purple sweet potato for 14 days. The water extract of purple sweet potato with a concentration ratio of 1:1
  Interventions: Other: The water extract of "Biang" variety purple sweet potato
- 1:6 water extract of purple sweet potato (Placebo Comparator): subjects were blindly and randomly assigned the lower concentration of water extract of purple sweet potato for 14 days. The water extract of purple sweet potato with a concentration ratio of 1:6
  Interventions: Other: The water extract of "Biang" variety purple sweet potato

INTERVENTIONS:
Other: The water extract of "Biang" variety purple sweet potato — Purple sweet potato extract is a mixture of water and "Biang" variety of purple sweet potato puree, enhanced with a touch of flavoring

SUMMARY:
Cerebral small vessel disease (CSVD) is a major cause of disability, cognitive impairment, and functional loss in the elderly. CSVD occurs due to damage to arterioles, capillaries, and venules in the brain parenchyma, and can cause clinical and neuroimaging symptoms. CSVD also accounts for up to 25% of all ischemic stroke cases, and making it the second leading cause of death in the world after ischemic heart disease.

Purple sweet potatoes, scientifically known as Ipomoea batatas (L.) Lam., contains of high anthocyanin specifically peonidin and cyanidin that has antioxidant, anti-inflammatory, and potentially phytoestrogenic activity. These anthocyanins have been linked to a reduced risk of obesity, diabetes, and high cholesterol. They also show potential in improving endothelial function, thereby enhancing blood vessel vasomotor function and potentially reducing the risk of cardiovascular diseases. Anthocyanins and their metabolites can cross the blood-brain barrier and affect signaling pathways, gene expression, and protein function at the molecular level. In addition to their ability to enhance vascular flow, anthocyanins can also help mitigate the risk factors associated with CSVD by counteracting oxidative stress in the body. These findings exploring the potential benefits of anthocyanins for individuals with CSVD by giving purple sweet potatoes extract comparing with placebo.

The outcomes that will be assessed are vasomotor reactivity measured by Breath Holding Index in Transcranial Doppler, Nitric Oxide, L-Arginine and Adiponectin levels in blood, Cognitive Test and Gait.

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the effectiveness of anthocyanins found in purple sweet potatoes as a functional food in individuals with CSVD. It is also hoped that anthocyanins could enhance the vasomotor reactivity of intracranial vessels in individuals with CSVD. Additionally, purple sweet potatoes may influence CSVD laboratory parameters, as well as functional gait and cognitive function.

The whole procedure will run for 16 days, divided into 3 parts (Pre-intervention, Intervention, and Post-intervention).

The participant will come in day 1 and 16. Pre-intervention (day 1) to conduct screening, provide informed consent, and also baseline assessment.

Intervention (day 2-15) involves consuming purple sweet potato extract (250 ml) twice daily, with daily delivery to maintain freshness. Additionally, patients will undergo a food recall assessment once on a weekday and twice on weekends.

Post-intervention (day 16) for continued outcome assessment.

The total number of visits from each participant is 2 times. The participant who meet the inclusion criteria and have signed the consent will be subjected to a baseline assessment followed by randomization into 2 groups/arms consisting of 2 treatments (1 group getting the water extract pf purple sweet potato) and 1 control group that got placebo. The daily food intake will be recorded by "3 days food diary-24 hours recall" method. The research team will contact the participant on 2 weekdays and 1 weekend day. The participant's regular medications will still be taken and recorded prior to the intervention.

Any unwanted event (adverse event) that occurs will be recorded. If an undesirable event occurs, a written report will be made to the ethics committee.

Demographic data will be presented descriptively according to the type of data. Univariate descriptive analysis will be used to provide an overview of the data. Data distribution test will be conducted using Kolmogorov-Smirnov. If the data is normally distributed, the t-test will be used, otherwise the Wilcoxon test will be used. Data analysis will be carried out using SPSS 25.0.

ELIGIBILITY:
Inclusion Criteria:

* CSVD patients aged 40-65 years.
* CSVD patients have been diagnosed by MRI.
* Willing to participate in the study and signed the consent letter after being given informed consent.
* Have a Montreal Cognitive Assessment score of at least 26.
* Able to walk independently with a motor score of at least 4, without proprioceptive disorders or neuropathy.

Exclusion Criteria:

* Closed temporal window on Transcranial Doppler examination
* Acute phase of stroke
* Hepatocellular injury
* Chronic kidney disease
* Intolerance to purple sweet potato
* Aphasia
* Neglected
* Visual impairment.
* Undergoing treatment with hormone replacement therapy (HRT), and corticosteroids.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Breath Holding Index | Through study completion, an average of 1 year
  The assessment will be conducted by a Neurologist who has special expertise in neurosonology using Transcranial Doppler.
  The outcome of this study is to find out the difference in scores from pre-intervention and post-intervention.
Nitric Oxide | Through study completion, an average of 1 year
  Nitric Oxide will be measured in plasma using Total Nitric Oxide and Nitrate/Nitrite Parameter Assay Kit.
  The outcome of this study is to find out the difference in concentration from pre-intervention and post-intervention.
L-Arginine | Through study completion, an average of 1 year
  L-arginine will be measured in plasma using L- Arginine Assay Kit (Colorimetry) The outcome of this study is to find out the difference in concentration from pre-intervention and post-intervention.
Adiponectin | Through study completion, an average of 1 year
  Adiponectin will be measured in serum using Human Total Adiponectin/Acrp30 Quantikine ELISA Kit The outcome of this study is to find out the difference in concentration from pre-intervention and post-intervention.
Cognitive | Through study completion, an average of 1 year
  The subjects will take a cognitive function test, namely Trail Making Test (TMT) A and Trail Making Test (TMT) B.
  The TMT-A test consists of combining numbers from 1 to 25, while the TMT-B test consists of alternating numbers and letters. TMT A and B are scored based on how long it takes to complete the test. This study is to find out the difference in scores from pre-intervention and post-intervention.
Gait | Through study completion, an average of 1 year
  The Timed Up and Go (TUG) test examination included assessment of the patient's balance, gait speed, and functional capacity. The TUG test assessment consisted of the subject standing up from a chair (chair height 46 cm, chair armrest height 65 cm), walking 3 meters, turning around, and walking 3-meters back to the chair and sitting down, at a spontaneous gait speed. The time taken to perform the test was measured using a stopwatch. The time recorded on the STANDARDIZED stopwatch was the TUG score.

CONTACTS AND LOCATIONS:
Overall Officials: Taufik Mesiano, MD, Principal Investigator — Doctoral Program in Medical Sciences Faculty of Medicine Universitas Indonesia

DOCUMENTS (1):
  • Informed Consent Form (2023-12-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT06380465/ICF_000.pdf